CLINICAL TRIAL: NCT04082546
Title: Correlates of Left Ventricular Global Longitudinal Strain and Surgical Intervention on Myocardial Bridges
Status: Completed | Type: Observational
Sponsor: ITAB - Institute for Advanced Biomedical Technologies (Other)
Collaborators: Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other)
Responsible Party: Principal Investigator, Francesco Bianco, Medical doctor, ITAB - Institute for Advanced Biomedical Technologies
Other Study IDs: CCPC001
Record Dates: First submitted 2019-09-03; First posted 2019-09-09 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Myocardial Bridge of Coronary Artery
Keywords: Coronary abnormalities; Angina; Global longitudinal strain; Speckle-traking echocardiography; Myocardial ischemia
MeSH Terms: conditions — Angina Pectoris; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical unroofing: Refractory angina to medical treatment (beta-blockers or calcium channels blockers)
  Interventions: Procedure: Surgical unroofing of muscle-briged coronary artery
- Medical treatment: Responders to medical treatment for angina relief
  Interventions: Procedure: Surgical unroofing of muscle-briged coronary artery

INTERVENTIONS:
Procedure: Surgical unroofing of muscle-briged coronary artery — Medical therapy with beta-blockers or calcium-channels blockers
  Other Names: Medical treatment

SUMMARY:
To examine the changes in left ventricular (LV) global longitudinal strain (GLS), using two-dimensional speckle tracking analysis, after left anterior descending (LAD) unroofing, in myocardial bridges (MBs) refractory to optimal medical therapy (OMT).

DETAILED DESCRIPTION:
The present study is enrolling all the MBs-patients who underwent angina surgical relief or medical treatment at the "Ospedali Riuniti" of Ancona, Italy, and the "University Hospital" of Chieti, Italy. All the participants will be examined utilizing echocardiography before and after the treatment. The two-dimensional speckle-tracking analysis will be performed with an off-line dedicated software from the apical 4-chambers-view. All the unroofing procedures will be performed under cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial bridge of the anterior descending left coronary artery

Exclusion Criteria:

* Poor echocardiographic imaging quality

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting a muscular myocardial bridge of the left anterior descending coronary artery causing chest discomfort/angina
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-11-26 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Improvement of myocardial function and contractility | 1 to 6 month after the procedure/treatment optimizzation
  The increment of global longitudinal strain analysis, from pre treatment values, as assessed by speckle-traking echocardiography

SECONDARY OUTCOMES:
Angina relief after surgical treatment | 1-month
  Defined as the reduction of CCS-Angina Scale, assessed by physicians, from grade I (ordinary physical activity does not cause angina, such as walking and climbing stairs) to grade IV (inability to carry on any physical activity without discomfort, anginal syndrome may be present at rest). The scale comprises 4 degrees in increasing order of angina severity.
Improvement in quality of life | 1-month
  Defined as the score increment, from 0 to 100 of the SAQ-7 questionnaire. The SAQ quantifies patients' physical limitations caused by angina, the frequency of and recent changes in their symptomstheir satisfaction with treatment, and the degree to which they perceive their disease to affect their quality of life. The questionnaire provides 7 different items with 6 different multiple choices. Each scale is transformed to a score of 0 to 100, where higher scores indicate better function (eg, less physical limitation, less angina, and better quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bianco, MD, Principal Investigator — G. d'Annunzio University
Locations (1):
- Ospedali Riuniti, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alegria JR, Herrmann J, Holmes DR Jr, Lerman A, Rihal CS. Myocardial bridging. Eur Heart J. 2005 Jun;26(12):1159-68. doi: 10.1093/eurheartj/ehi203. Epub 2005 Mar 11. PMID 15764618
- [Background] Corban MT, Hung OY, Eshtehardi P, Rasoul-Arzrumly E, McDaniel M, Mekonnen G, Timmins LH, Lutz J, Guyton RA, Samady H. Myocardial bridging: contemporary understanding of pathophysiology with implications for diagnostic and therapeutic strategies. J Am Coll Cardiol. 2014 Jun 10;63(22):2346-2355. doi: 10.1016/j.jacc.2014.01.049. Epub 2014 Feb 26. PMID 24583304
- [Background] Cerit L, Duygu H. Myocardial bridging and sudden death. Int J Cardiol. 2017 Feb 15;229:11. doi: 10.1016/j.ijcard.2016.11.308. Epub 2016 Dec 1. No abstract available. PMID 27923515
- [Background] Zhang M, Yang J, Ma C, Liu M. Longitudinal strain measured by two-dimensional speckle tracking echocardiography to evaluate left ventricular function in patients with myocardial bridging of the left anterior descending coronary artery. Echocardiography. 2019 Jun;36(6):1066-1073. doi: 10.1111/echo.14357. Epub 2019 May 13. PMID 31087389
- [Background] Alessandri N, Dei Giudici A, De Angelis S, Urciuoli F, Garante MC, Di Matteo A. Efficacy of calcium channel blockers in the treatment of the myocardial bridging: a pilot study. Eur Rev Med Pharmacol Sci. 2012 Jun;16(6):829-34. PMID 22913217